CLINICAL TRIAL: NCT05686499
Title: Building Capacity for Screening & Early Diagnosis of Colorectal Cancer Through a Comprehensive Colonoscopy Training Program in Nigeria
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Obafemi Awolowo University Teaching Hospital (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Principal Investigator, Olusegun Alatise, professor, Obafemi Awolowo University Teaching Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ERC/2022/07/03
Record Dates: First submitted 2022-07-25; First posted 2023-01-17 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Trainees will be selected from among resident doctors and consultants working in teaching hospitals and federal medical centres that have facilities for colonoscopy. These will be randomized into two arms - high fidelity (HF) and low fidelity (LF) arms. Baseline test will then be carried out by the trainees after which they will be exposed to colonoscopy lectures and demonstrations using respective fidelity type to which they are randomized. Simulation examination will then be carried out after which trainees will be cross-overed to alternate arms for further simulation on different fidelity types. They will then all have opportunity to perform colonoscopy on live patients which will be supervised and accessed by trainers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Fidelity (HF) Arm (Active Comparator): The HF simulator will be Limbs and Things Colonoscopy Training Model product KKM40.
  Interventions: Other: Didactic Lectures and demonstrations
- Low Fidelity (LF) Arm (Experimental): The LF simulator will be made in Nigeria, based on low fidelity models that have been published in the literature
  Interventions: Other: Didactic Lectures and demonstrations

INTERVENTIONS:
Other: Didactic Lectures and demonstrations — 1. Trainees will receive 4-6 hours of didactic colonscopy lecture sessions based on the American Board of Surgery Flexible Endoscopy curriculum for general surgery residents, general surgery resident curriculum (SCORE) endoscopy module, and the Joint Advisory group on GI Endoscopy program adapted to Nigeria context.
  2. Trainees will have the opportunity to practice colonoscopy on HF or LF simulators (depending on the arm) with immediate feedback from instructors.

SUMMARY:
This protocol seeks to develop a colonoscopy training program in Nigeria in order to increase the number of health care providers proficient in colonoscopy. The goal is to improve capacity for screening and early diagnosis of colorectal cancer (CRC) by training and expanding the healthcare workforce that is competent in endoscopy techniques. The project has three components, a needs assessment, simulation training, and training on live patients.

The first part of this project determines the number of providers and endoscopy procedures currently performed in Nigeria, as well as patient access to facilities that have colonoscopy capabilities, through a mixed methods approach. Surveys, focus in-depth interviews with key stakeholders, and use geographic information system (GIS) modeling technology will be employed to perform a needs assessment. The second component of this project investigates whether a locally developed low fidelity (LF) simulation colonoscopy training model is an effective teaching, training, and assessment tool for skill acquisition and confidence compared to a high-fidelity (HF) colonoscopy model. The third component of this project is training healthcare providers on real patients who have an indication for colonoscopy. This project seeks to build capacity for endoscopy services in order to increase capacity for screening and early diagnosis of CRC. At the end of the project, it is expected the number of providers trained to perform colonoscopy in a resource limited setting like Nigeria will increase.

DETAILED DESCRIPTION:
The goal of this project is to build capacity for early diagnosis of CRC by developing a comprehensive colonoscopy training program that could in the future lead to credentialing and accreditation of a trainee. The first aspect of the project focuses on needs assessment analysis as it determines the quantity of providers and access to facilities that perform colonoscopy through surveys, focus in-depth interviews, and GIS technology. The second component investigates whether a locally developed LF simulation colonoscopy training tool is an effective teaching, training, and assessment tool for skill acquisition and confidence compared to a HF colonoscopy model in a resource limited setting. The third component of the project will assess whether training on a low or high-fidelity simulator then translates to improved performance of colonoscopy on live patients. At the end of the project, it is expected the number of providers trained to perform colonoscopy in a resource limited setting like Nigeria will increase.

OVERVIEW OF STUDY DESIGN/INTERVENTION A mixed methods survey was developed that determines the baseline number of endoscopists, nurses, anaesthetists, ancillary staff, costs, and the number of procedures performed per year in endoscopy centers in the country of Nigeria. This survey will be developed with qualitative specialists at the Obafemi Awolowo University (OAU) and the Memorial Sloan Kettering Cancer Center (MSKCC). Healthcare professionals who are part of Nigerian medical societies will be invited to participate in the survey through paper, electronic, or social media platforms. Focused in-depth interviews with key stakeholders will be conducted to further understand the barriers to endoscopy care in Nigeria.

Prior to participating in this survey study, the purpose of the study will be explained to potential participants. They will be provided information about the research study in written form and a consent form will be provided. Consent will be obtained in written form in English, since this is the national language medium used for medical professionals in Nigeria.

Results from this survey and collaborations with medical societies in Nigeria, will provide information needed to identify which healthcare facilities perform endoscopy in Nigeria. GIS technology will be utilized to analyze patient access to these facilities based on locations of facilities to neighborhoods where patients may reside. Qualitative surveys and focus interviews with key stakeholders will also provide information on barriers to accessing and providing care to patients who need colonoscopy.

For the simulation training portion of the study, following initial recruitment, an equal number of consented participants will be randomized to learn colonoscopy on high or low fidelity models. The HF simulator will be Limbs and Things Colonoscopy Training Model product KKM40. The LF simulator will be made in Nigeria, based on low fidelity models that have been published in the literature. Prior to beginning the course, the participants will be given instructions, a prior experience and confidence survey, and then will be asked to perform colonoscopy. This first assessment will serve as a baseline measure of colonoscopy skills. The LF group will perform a pretest on LF models, and the HF group will perform the pre-test on HF models. Participants will be evaluated utilizing the Mayo colonoscopy skills assessment tool and the Global Assessment of Gastrointestinal Endoscopic Skills (GAGES) tools that have been validated and published in the literature previously.

Following this pre-test, study participants will partake in didactic teaching sessions. The colonoscopy lecture curriculum will be adapted for the Nigerian context and standardized utilizing content based on the American Board of Surgery Flexible Endoscopy curriculum for general surgery residents, general surgery resident curriculum (SCORE) endoscopy module, and the Joint Advisory group on GI Endoscopy program. Teaching sessions between high and low fidelity groups will be identical except for the type of simulation models used to demonstrate and practice colonoscopy. Trainees will have the opportunity to practice colonoscopy on simulators with immediate feedback from instructors.

After this 4-6-hour teaching session, participants will take a post-test identical to the colonoscopy pre-test. The next day participants will perform colonoscopy procedures on live patients and be evaluated on live patients utilizing the GAGES and mayo colonoscopy skills assessment tools. Additionally, at the end of the study, participants will be asked to fill out a confidence survey During the live patient sessions, the study will involve patients who were scheduled to undergo a clinically indicated colonoscopy. The patients will sign a consent form to be part of the study which allows trainees to perform colonoscopy under the direct supervision by trained colonoscopy physician. The trainee will be the primary endoscopist under the supervision of a faculty endoscopy evaluator. The evaluator will allow the study participants independence while ensuring patient safety. The instructor can provide verbal instruction if necessary. If the instructors feel the study participant is not making progress or if patient safety is of concern, the instructors are permitted to take control of the colonoscopy and navigate through difficult portions of the colon or takeover the procedure completely. The maximum time that will be allotted for the trainee to complete the colonoscopy will be 30 minutes. A critical flaw point will be given to the trainee participant if complete takeover occurs, although they will be given the opportunity to try again on a different patient if feasible.

Trainees will also be evaluated based on total procedure time, time to rectosigmoid junction, splenic flexure, hepatic flexure and cecal intubation, % of successful cecal intubation, % of time for which the view of the lumen was lost, % of times TI intubation successful, and withdrawal time of colonoscopy from cecum, avoidance of bowel perforation and median depth of maximal insertion based on the following scale: 1 = rectum, 2 = sigmoid, 3 = descending colon, 4 = splenic flexure, 5 = transverse colon, 6 = hepatic flexure, 7 = ascending colon, 8 = cecum. Additionally, at the end of the study, participants will be asked to fill out course satisfaction and confidence surveys.

PRIMARY AND SECONDARY OUTCOMES Primary Outcome: To determine whether learning colonoscopy on a LF simulation model confers similar skill acquisition and confidence as training on a HF model Secondary Outcomes: Determine access to endoscopists and endoscopy facilities barriers to endoscopy, and costs of endoscopy in Nigeria. Assess whether training on a low or high-fidelity simulator improves colonoscopy performance on real patients. To evaluate the overall improvement in technical skills of trainees before and after delivery of a simulation-based colonoscopy training program designed to teach colonoscopy in a resource limited setting. Investigators will also determine costs of implementing a colonoscopy training program as well as costs of endoscopy at each of the facilities.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Health care professionals will include consultants and registrars in medicine, surgery, and gastroenterology

Exclusion Criteria:

* Participants under the age of 18
* Participants unwilling to sign consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
ratio of low-fidelity simulator trained endoscopists with improved colonoscopy performance on real patients to high-fidelity simulator trained endoscopists with improved performance on real patients | 5 days
  proportion of LF simulator training who can perform colonoscopy adequately on live patient to proportion of HF simulator training who can perform colonoscopy adequately on live patients

CONTACTS AND LOCATIONS:
Locations (2):
- Nigeria (2):
  - Endoscopy Unit, Obafemi Awolowo University Teaching Hospitals, Ile-Ife, Osun State
  - Obafemi Awolowo University Teaching Hospitals Complex, Ile-Ife, Osun State

IPD SHARING:
Plan to Share IPD: Yes
There is an existing collaboration betweeen OAUTHC and MSKCC. The current data transfer agreement will be amended to include this specific protocol. Data will be collected on redcap and be de-identified at the point of analysis
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available within three months of study commencement and it will be hosted on the redcap for 10years
Access Criteria: Being a research staff (principal investigator, co-investigators, programme / clinical research managers, clinical research coordinators, research assistants) working in the two collaborative sites